CLINICAL TRIAL: NCT05224557
Title: Analysis of Cardiac Biomarker Racial Discrepancies in African American Patients With Heart Failure With Reduced Ejection Fraction
Brief Title: Analysis of Cardiac Biomarker Racial Discrepancies
Status: Enrolling by invitation | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 043.PHA.2021.A
Record Dates: First submitted 2022-02-03; First posted 2022-02-04 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- New onset HFrEF AA patients: New onset HFrEF AA patients
  Interventions: Other: No intervention
- New onset HFrEF Caucasian patients: New onset HFrEF Caucasian patients
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The goal is to review cardiac biomarkers present on admission between African American patients with new onset Heart Failure compared to a comparable cohort of Caucasian patients to establish whether there is a clinically significant difference between the two groups regarding cardiac biomarker levels and initial Heart Failure severity.

Hypothesis: Cardiac biomarker levels in African American patients with new onset Heart Failure with Reduced Ejection Fraction will be significantly lower than a Caucasian cohort with new onset Heart Failure with Reduced Ejection Fraction.

DETAILED DESCRIPTION:
Limited data exists on the overall impact racial and genetic differences play on expression of cardiac biomarkers, especially natriuretic peptides (NPs). NPs like atrial NP, brain NP (BNP), and C-type NP are endogenous hormones with powerful cardiovascular and metabolic effects. NPs play an active role in natriuresis and vasodilation along with lipolysis, weight loss, and insulin sensitivity, whereas NP deficiencies correlate with increased risk for developing cardiovascular comorbidities like hypertension. Many cardiac disease states like acute coronary syndrome, valvular heart disease (VHD), and atrial fibrillation (AFib) can cause significant elevations in NPs. Elevated NP levels have also been associated with liver cirrhosis, chronic renal dysfunction, and infectious sepsis. However, NP elevations are most commonly associated with heart failure (HF), and increasing BNP levels have been correlated with increasing grades of cardiac dysfunction and end-diastolic wall stress within the heart.

African American (AA) patients experience higher incidence of HF relative to the general population and are at an increased risk of mortality secondary to chronic HF compared to Caucasian patients. AA patients are three times more likely to develop HF because AA patients may suffer from a subgroup of left ventricular hypertrophy where biomarkers like N-terminal pro-BNP (NT-proBNP) are not clinically elevated. The 2021 American College of Cardiology/American Heart Association Heart Failure with Reduced Ejection Fraction (HFrEF) Treatment Guidelines endorse measurement of both BNP and NT-proBNP as biomarkers for the diagnosis and prognostication of HF; however, current treatment guidelines have not established treatment thresholds for either BNP or NT-proBNP.7 The Food and Drug Administration (FDA) approved cutoff BNP value for the diagnosis of HF is 100 pg/mL. For NT-proBNP, the optimal cutoff values for confirmatory decision limits for HF are 450, 900, and 1,800 pg/mL for ages less than 50 years, between 50 to 75 years, and older than 75 years of age, respectively.3 In clinical practice, significant heterogeneity surrounds treatment cutoffs for NT-proBNP levels for treatment of HF, as seen in many recent prominent landmark HF pharmacotherapy trials.

Within the general population, serum NP levels, especially NT-proBNP, are significantly lower in the AA population compared to Caucasians as seen in the Reasons for Geographic and Racial Differences in Stroke, Dallas Heart, and Atherosclerosis Risk in Communities studies. After accounting for traditional risk factors, racial differences in body composition, cardiac structure, and socioeconomic factors, AA patients were found to have significantly lower serum NT-proBNP levels and greater levels of markers of myocardial stress and inflammation, including high-sensitivity Troponin T (hsTnT), GDF-15, and ST2. This finding may also be due to genetic differences, as percent European ancestry (PEA) in AA patients was found to have a direct impact on NT-proBNP levels in the general AA population. Of the 1656 AA patients in whom PEA data were available, a 10% increase in PEA was associated with 7% higher adjusted NT-proBNP levels.

Knowing that the general AA population has lower serum NP's compared to Caucasian patients, limited research focuses on initial NT-proBNP levels in AA patients with new-onset HF. Given that many landmark HF trials primarily enroll Caucasian patients, several questions emerge: (i) should medicine individualize treatment thresholds for NT-proBNP and other cardiac biomarkers based on race given known racial discrepancies with serum NP's and increased mortality seen in these patients? (ii) Is the trend seen in AA patients regarding serum NPs and other cardiac biomarkers still true when these patients present with new-onset HF? Our goal is to review cardiac biomarkers present on admission between AA patients with new onset HF compared to a comparable cohort of Caucasian patients to establish whether there is a clinically significant difference between the two groups regarding cardiac biomarker levels and initial HF severity.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* Self-identified as AA
* Self-identified as Caucasian
* NYHA class II-IV symptoms
* Left ventricle EF <40%
* First admission for HFrEF
* No echocardiography during initial admission

Exclusion Criteria:

* Patients not meeting inclusion criteria

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects that self-identify as African American or Caucasian with a new onset of Heart Failure with Reduced Ejection Fraction
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2024-08-15 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
Baseline NT-proBNP levels on admission | Chart reviews ill be done for charts generated from April 2017 to August 2020
  Collection of baseline blood tests
Baseline troponin-I or troponin-T levels on admission | Chart reviews ill be done for charts generated from April 2017 to August 2020
  Collection of baseline blood tests
Demographic data: Age | Chart reviews ill be done for charts generated from April 2017 to August 2020
  Age of subject in years
Demographic data: Gender | Chart reviews ill be done for charts generated from April 2017 to August 2020
  male or female
Demographic data: body mass index (BMI) | Chart reviews ill be done for charts generated from April 2017 to August 2020
  BMI is calculated by taking the weight in kilograms divided by height in meters squared
Ejection Fraction on echocardiography during first admission | Chart reviews ill be done for charts generated from April 2017 to August 2020
  The patient has an EF <40% on echocardiography and is not on goal-directed medical therapy for HFrEF.
New York Heart Association (NYHA) class | Chart reviews ill be done for charts generated from April 2017 to August 2020
  Doctors usually classify patients' heart failure according to the severity of their symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Crystal Brown, PharmD, Principal Investigator — Methodist Health System
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No